CLINICAL TRIAL: NCT02011906
Title: The Effects of Omega 3 and Vitamin E Supplementation on the Serum Antioxidant Enzymes and Gene Expressions of PGC-1a, h TERT, FOXOs and SIRTs in CAD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95983
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: antioxidant enzymes; omega 3; vitamin E; CAD; Sirtuins; FOXOs
MeSH Terms: conditions — Coronary Artery Disease | interventions — Docosahexaenoic Acids; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CAD, OMEGA 3 (Active Comparator): patients with CAD who receive 4 gr/day omega 3 in the form of 4 softgels each of them contains 1000 mg omega 3 and a softgel contains placebo of vitamin E
  Interventions: Dietary Supplement: omega 3; Dietary Supplement: placebo of vitamin E
- CAD, omega 3 and vitamin E (Active Comparator): patients with CAD who receive 4 gr/day omega 3 in the form of 4 softgels each of them contains 1000 mg omega 3 and a softgel contains 400 IU vitamin E
  Interventions: Dietary Supplement: omega 3; Dietary Supplement: vitamin E
- CAD, placebo (Placebo Comparator): patients with CAD who receive 4 softgels/day each of them contains placebo of omega 3 and a softgel/day contains placebo of vitamin E
  Interventions: Dietary Supplement: placebo of omega 3; Dietary Supplement: placebo of vitamin E

INTERVENTIONS:
Dietary Supplement: omega 3
  Arms: CAD, OMEGA 3; CAD, omega 3 and vitamin E
Dietary Supplement: vitamin E
  Arms: CAD, omega 3 and vitamin E
Dietary Supplement: placebo of omega 3
  Arms: CAD, placebo
Dietary Supplement: placebo of vitamin E
  Arms: CAD, OMEGA 3; CAD, placebo

SUMMARY:
The aim of this study is to determine the effects of omega 3 supplementation and its concurrent supplementation with vitamin E on the serum levels of antioxidant enzymes and the expressions of the PGC-1a, h TERT, FOXO1, FOXO3a , SIRT1,SIRT3, SIRT6 genes in PBMC cells in the patients with coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

-

literate, willingness to participation, CAD patients 45- 65 years old, body mass index< 30, avoidance of dietary supplements, vitamins and herbal products at least 3 months before and throughout the intervention, willing to maintain body weight during the study

Exclusion Criteria:

* people who have used vitamin E or omega 3 supplements in last 3 months, having chronic renal disease ,cancer, Hepatobilliary diseases, hematological disorders, hypo- or hyperthyroidism, diabetes, treatment with PPAR-gamma agonists or Thiazolidinediones, Smokers

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
serum total cholesterol | change from baseline at 2 months
serum HDL cholesterol | change from baseline at 2 months
serum triglycerides level | change from baseline at 2 months
serum LDL cholesterol | change from baseline at 2 months
serum insulin | change from baseline at 2 months
serum Hs-CRP | change from baseline at 2 months
serum gluthatione peroxidase | change from baseline at 2 months
serum catalase | change from baseline at 2 months
serum superoxide dismutase | change from baseline at 2 months
serum total antioxidant capacity | change from baseline at 2 months

SECONDARY OUTCOMES:
gene expression of SIRT1 | change from baseline at 2 months
gene expression of SIRT3 | change from baseline at 2 months
gene expression of SIRT6 | change from baseline at 2 months
gene expression of PGC-1a | change from baseline at 2 months
gene expression of FOXO3a | change from baseline at 2 months
gene expression of FOXO1 | change from baseline at 2 months
gene expression of h TERT | change from baseline at 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran